CLINICAL TRIAL: NCT07346092
Title: Health Perceptions and Social Behaviors in Young Adults
Brief Title: Studying the Health Perceptions and Social Behaviors of Graduate Students at the Ohio State University for the Development of Effective Oral Nicotine Pouch Addictive Risk Communication
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Megan Roberts, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OSU-24421; NCI-2025-07731 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); U54CA287392 (NIH)
Record Dates: First submitted 2025-12-29; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Tobacco-Related Carcinoma

STUDY DESIGN:
Intervention Model Description: Students identified in Aim 1 as susceptible to ONPs, having experimented with ONPs, or currently using ONPs will be invited to participate in Aim 2 or Aim 3. In Aim 2, participants will view four randomly selected messages from the five message blocks and complete brief evaluations after each message. In Aim 3, participants who consent will be randomly assigned to view either static or dynamic visual ONP risk messages.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Aim 1 (online survey) (No Intervention): Participants complete an online survey assessing ONP use patterns, perceptions of ONP-related norms, and interactions with ONP content on social media over 5-10 minutes on study.
- Aim 2 (Experimental): Participants view four intervention messages shown in a randomized order. These messages are randomly selected from five message blocks, which are part of a total pool of 33 messages.
  Interventions: Other: Preventive Intervention; Other: Survey Administration
- Aim 3 condition I (static visual ONP risk messages) (Active Comparator): Participants view static visual ONP risk messages on study.
  Interventions: Other: Preventive Intervention; Other: Survey Administration
- Aim 3 condition II (dynamic visual ONP risk messages) (Experimental): Participants view dynamic visual ONP risk messages on study.
  Interventions: Other: Preventive Intervention; Other: Survey Administration

INTERVENTIONS:
Other: Preventive Intervention — View social norm-based ONP messages
  Other Names: PREVENTATIVE; Prevention; Prevention Measures; Prophylactic; Prophylaxis; PRYLX
  Arms: Aim 2
Other: Preventive Intervention — View static visual ONP risk messages
  Other Names: PREVENTATIVE; Prevention; Prevention Measures; Prophylactic; Prophylaxis; PRYLX
  Arms: Aim 3 condition I (static visual ONP risk messages)
Other: Preventive Intervention — View dynamic visual ONP risk messages
  Other Names: PREVENTATIVE; Prevention; Prevention Measures; Prophylactic; Prophylaxis; PRYLX
  Arms: Aim 3 condition II (dynamic visual ONP risk messages)
Other: Survey Administration — Ancillary studies
  Arms: Aim 2; Aim 3 condition I (static visual ONP risk messages); Aim 3 condition II (dynamic visual ONP risk messages)

SUMMARY:
This clinical trial studies the health perceptions and social behaviors of Ohio State University (OSU) graduate students to develop an interactive, social norms-based approach that is effective in communicating the addictive risks of oral nicotine pouches (ONPs). The use of ONPs is rising rapidly among young adults (YA). Various factors contribute to the growing popularity of ONPs, including their affordability, accessibility both online and in physical stores, discreet use, and heavy internet advertising. However, for those who are experimenting, have tried ONPs in the past, or have never used them but are surrounded by others who do, factors like affordability and availability may not be the only reasons for initiating or continuing use. Social norms are also a significant factor influencing YA tobacco use. Peer influence on college campuses and in other social environments may encourage YA to conform to behaviors they perceive as popular or acceptable. Being surrounded by peers who use ONPs may create pressure to try them, especially as YA seek to fit in within their social circles. Studying the health perceptions and social behaviors of OSU graduate students may help researchers develop an interactive, social norms-based approach that is effective in communicating the addictive risks of ONPs.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate OSU graduate students' ONP use patterns, perceptions of use within their social circles, and ONP information-gathering behaviors on social media.

II. Test the effects of normative-focused, YA-directed ONP risk messages to enhance knowledge and correct misperceptions about addiction.

III. Estimate the effect of dynamic versus (vs.) static visual ONP risk messages on YA's information-sharing intentions.

OUTLINE: All participants will first complete Aim 1. Participants identified as high risk for nicotine dependence and who consent to follow up will then be randomly assigned to Aim 2 or Aim 3.

AIM 1: Participants complete an online survey assessing ONP use patterns, perceptions of ONP-related norms, and interactions with ONP content on social media over 5-10 minutes on study.

AIM 2: Participants view four intervention messages shown in a randomized order. These messages are randomly selected from five message blocks, which are part of a total pool of 33 messages. After viewing each message, participants complete a brief questionnaire that assesses perceived message effectiveness, ONP-related knowledge, risk perceptions, and self-efficacy.

AIM 3: Participants are randomly assigned to 1 of 2 conditions.

CONDITION I: Participants view static visual ONP risk messages on study.

CONDITION II: Participants view dynamic visual ONP risk messages on study.

Following message exposure, participants will answer questions about their intentions to use ONPs in the future, perceived susceptibility, beliefs, attitudes toward ONPs, and cognitive responses (e.g., perceived message effectiveness).

ELIGIBILITY:
Inclusion Criteria:

* AIM 1: OSU graduate students aged 21 years or older
* AIM 2 AND 3: Students identified in Aim 1 as susceptible to ONPs, having experimented with ONPs, or currently using ONPs-those considered at high risk for nicotine dependence-will be invited to participate in Aim 2 or Aim 3
* AIM 3: Participants in Aim 2 will not be invited to participate in Aim 3, as they will have already been exposed to the experimental stimuli

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2027-03-20 (Estimated); Study Completion 2027-03-20 (Estimated)

PRIMARY OUTCOMES:
Susceptibility to Oral Nicotine Pouch (ONP) Use (Three Item Susceptibility Scale) (Aim 1) | Up to 2 years
  Susceptibility will be measured using three validated items assessing the likelihood of trying ONPs in the future (e.g., "Would you try an ONP if offered by a friend?"). Responses will be scored on a Likert scale and averaged to form a composite susceptibility index.
ONP Related Perceptions (Multi-Item Perception Scales) (Aim 1) | Up to 2 years
  Participants will rate perceived harm and comparative risks of ONPs using validated scales. Responses will be scored on a Likert scale and averaged to form a composite perception index.
Normative Perceptions of ONP Use (Descriptive, Injunctive, Subjective Norm Scales) (Aim 1) | Up to 2 years
  Participants will report perceived prevalence of ONP use among peers, perceived approval or disapproval from important others, and perceived expectations regarding ONP use. Scale scores will be computed for each norm type.
Exposure to ONP Information on Social Media (Self Report Communication Channel Checklist) (Aim 1) | up to 2 years
  Participants will indicate which social media platforms and communication channels they encounter ONP related content on, and frequency of exposure.
ONP Risk Perceptions (Risk Perception Items) (Aim 2, Aim 3) | Up to 2 years
  Participants will rate perceived likelihood and severity of harms associated with ONP use using validated risk perception scales.
Self Efficacy to Avoid ONP Use (Self Efficacy Scale) (Aim 2, Aim 3) | Up to 2 years
  Self-efficacy will be measured using items assessing confidence in avoiding ONP use in tempting or high-risk situations. Scores will be averaged to create a self efficacy index.
Perceived Message Effectiveness (PME Scale) (Aim 2, Aim 3) | up to 2 years
  After each message, participants will complete a validated perceived message effectiveness scale assessing attention, relevance, and persuasiveness. Scores will be aggregated per message.
Intentions to share on social media (Intention Scale)(Aim 3) | Up to 2 years
  Participants will rate the likelihood of sharing the information about ONP messages on social media using validated intention items. Responses will be averaged into a composite intention score.
Attitudes Toward ONPs (Attitudinal Scales) (Aim 3) | up to 2 years
  Participants will complete validated scales measuring cognitive and affective attitudes toward ONPs. Scale totals or means will serve as outcome metrics.
Cognitive Responses to Message Exposure (Message Response Items) (Aim 3) | up to 2 years
  Participants will rate message clarity, believability, engagement, and perceived effectiveness using validated cognitive response items.

SECONDARY OUTCOMES:
Tobacco Use History (Self Report Questionnaire) (Aim 1) | up to 2 years
  Participants will report past and current use of tobacco products, including oral nicotine pouches (ONPs) and other tobacco/nicotine products. Data will include categorical indicators of ever use, past 30 day use, frequency, and product types.
Sociodemographic Characteristics (Aim 1, Aim 2, Aim 3) | up to 2 years
  Participants will provide demographic data, including age, gender, race/ethnicity, educational program, and other demographic characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Megan E Roberts, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu